CLINICAL TRIAL: NCT00667069
Title: Randomized, Multicenter Study Comparing the Immediate Adjuvant Radiotherapy Associate With Hormonal Therapy of LH-RH Analogue (Decapeptyl® LP) vs Delayed Radiotherapy Until Biochemical Relapse Associated With Hormonal Therapy of LH-RH Analogue (Decapeptyl® LP) in Patients With Operable Prostate Cancer pT3 R1 pN0 or pNx at Intermediate Risk.
Brief Title: Triptorelin and Radiation Therapy in Treating Patients Who Have Undergone Surgery for Intermediate-Risk Stage III or Stage IV Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU 17 - UC-0160/0702; 2007-002495-34 (EudraCT Number); CDR0000577485 (Other: Unicancer)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Chemotherapy, Adjuvant; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Relapse (Other): Radiotherapy and Hormonotherapy only if relapse
  Interventions: Drug: triptorelin; Procedure: adjuvant therapy; Radiation: 3-dimensional conformal radiation therapy
- B Immediate treatment (Experimental): Radiotherapy and Hormonotherapy at randomization
  Interventions: Drug: triptorelin; Procedure: adjuvant therapy; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Drug: triptorelin
  Other Names: Decapeptyl
Procedure: adjuvant therapy
Radiation: 3-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as triptorelin, may lessen the amount of androgens made by the body. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether giving triptorelin and radiation therapy soon after surgery or later after surgery is more effective in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying giving triptorelin and radiation therapy soon after surgery to see how well it works compared with giving them later after surgery in treating patients who have undergone surgery for intermediate-risk stage III or stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy, in terms of event-free survival at 5 years, of immediate radio-hormonal therapy immediately after prostatectomy for tumor pT2, R1, pN0, or pNx versus radio-hormonal therapy at biochemical relapse.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the metastasis-free survival of these patients.
* Compare the acute and late toxicities of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the functional dependence of patients over 75 years old.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I (delayed treatment): Patients receive triptorelin intramuscularly on day 1 and then 3 months later. Patients also undergo conformal radiotherapy daily, 5 days a week, for 7 weeks. Treatment begins at biochemical relapse (PSA is more than 0.2 ng/mL) and before PSA is more than 2 ng/mL.
* Arm II (immediate treatment): Patients receive treatment as in arm I, but treatment begins within 6 months after surgery.

After completion of study treatment, patients are followed for up to 5 years.

ELIGIBILITY:
Inclusion criteria:

1. Patient must have undergone curative surgery for a localized adenocarcinoma of the prostate
2. pT3a, pT3b (or pT4 by reaching the bladder neck), or R1 disease (stage III or IV)
3. PSA ≤0.1 ng/mL after prostatectomy (confirmed at 1 month)
4. May receive treatment within 6 months after surgery
5. Positive margins (tumoral glands in contact with contour ink) on the surgical specimen
6. pN0 or pNx (lymph nodes resected during negative prostatectomy or lymph nodes not resected)
7. No current clinical or biochemical progressive disease
8. Life expectancy ≥10 years
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
10. Patient must be affiliated to the social security system
11. Patient must have received the information sheet and signed the consent form

Exclusion criteria:

1. Patient with prostate cancer other than adenocarcinoma
2. Gleason score ≥8 and with seminal vesicles involved
3. pN1 disease (Histologically confirmed nodal invasion during initial lymph node resection)
4. pT2 disease
5. Prior surgical or chemical castration
6. Prior hormonal therapy
7. Prior radiotherapy within 3 months after radical prostatectomy
8. Prior pelvic radiotherapy
9. No history of cancer (except basal cell skin cancer) within 5 years of surgery
10. No known severe hypertension uncontrolled by appropriate therapy (≥160 mm Hg systolic and/or ≥90 mm Hg diastolic)
11. Known hypersensitivity to gonadotropin-releasing hormone or its analogs
12. Contraindication to intramuscular injection
13. Concurrent participation in another interventional study
14. Patients under protective custody or guardianship, unable to comply with the specific requirements of the study or unable to understand the purpose of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2008-04-07 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Event-free survival | From randomization to disease progression or death, up to 5 years
  The event-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse (clinical progression, biochemical progression, death)

SECONDARY OUTCOMES:
Overall survival | From randomization to death from any cause, up to 10 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Metastases-free survival | From randomization to metastases onset, up to 10 years
  The metastases-free survival is the length of time during and after the treatment for cancer that a patient is still alive and the cancer has not spread to other parts of the body.
Acute or chronic toxicity | Throughout study completion, up to 10 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 3 (NCI-CTCAE v3.0) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale will assess the severity of sensory neuropathic disorders, this derivative into 5 grades determined by the investigator.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 2 years, and 5 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Prostate Cancer Module (QLQ-PR25) | At baseline, 2 years, and 5 years
  This EORTC prostate cancer specific questionnaire is intended to supplement the QLQ-C30.
  The prostate cancer module is a 25-item questionnaire designed for use among patients with localized and metastatic prostate cancer. It includes subscales assessing urinary symptoms (9 items), bowel symptoms (4 items), treatment-related symptoms (6 items), and sexual functioning (6 items). Using a 4-point Likert scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), patients indicate the degree to which they have experienced symptoms.
Functional dependence in patients over 75 years old | At baseline, 2 years, and 5 years
  The Lawton Instrumental Activities of Daily Living (IADL) Scale is a self-reported questionnaire to assess independent living skills for older adults. This questionnaire, composed of 31 questions organized into 8 domains (ability to use telephone, shopping, food preparation, housekeeping, laundering, mode of transportation, responsibility for own medications, and ability to handle finances), is designed to identify improvement or deterioration of a person functioning over time. Each domain is scored 0-1 for a summary score ranging from 0 (low function, dependent) to 8 (high function, independent).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Richaud, MD, Study Chair — Institut Bergonié
Locations (17):
- France (17):
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Hopitaux Civils de Colmar, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Leon Berard, Lyon
  - Clinique du Pont de Chaume, Montauban
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Centre Henri Becquerel, Rouen
  - Centre Regional Rene Gauducheau, Saint-Herblain
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sargos P, Chabaud S, Latorzeff I, Magne N, Benyoucef A, Supiot S, Pasquier D, Abdiche MS, Gilliot O, Graff-Cailleaud P, Silva M, Bergerot P, Baumann P, Belkacemi Y, Azria D, Brihoum M, Soulie M, Richaud P. Adjuvant radiotherapy versus early salvage radiotherapy plus short-term androgen deprivation therapy in men with localised prostate cancer after radical prostatectomy (GETUG-AFU 17): a randomised, phase 3 trial. Lancet Oncol. 2020 Oct;21(10):1341-1352. doi: 10.1016/S1470-2045(20)30454-X. PMID 33002438
- [Derived] Campillo-Gimenez B, Buscail C, Zekri O, Laguerre B, Le Prise E, De Crevoisier R, Cuggia M. Improving the pre-screening of eligible patients in order to increase enrollment in cancer clinical trials. Trials. 2015 Jan 16;16:15. doi: 10.1186/s13063-014-0535-7. PMID 25592642